CLINICAL TRIAL: NCT05127603
Title: The Effect of Cognition Targeted Physical Therapy in People With Non-specific Neck Pain: A Mixed-Method Multiple Case Study
Brief Title: The Effect of Cognition Targeted Physical Therapy in People With Non-specific Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rotterdam University of Applied Sciences (Other)
Collaborators: VU University of Amsterdam (Other); Multiple primary care physical therapy clinics (Unknown)
Responsible Party: Principal Investigator, Maaike Kragting, Principal Investigator, PhD-student, Physical Therapist and Lecturer, Rotterdam University of Applied Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR01_MCS_NeckPain
Record Dates: First submitted 2021-11-01; First posted 2021-11-19 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Neck Pain
Keywords: Pain; Psychological Intervention; Qualitative evaluation; Quantitative evaluation
MeSH Terms: conditions — Neck Pain; Pain

STUDY DESIGN:
Intervention Model Description: Single Case methodology with a baseline (phase A), intervention (phase B) and intervention withdrawal phase (A')
  This multiple case study has three phases: (A) A baseline phase of two weeks with no intervention, (B) a treatment phase with 5-7 consultations (offered weekly) and (A') a follow-up 3 months after the last treatment consultation.
  The participants are seen as single systems in both the qualitative as the quantitative analyses in an experimental design, using a tailored care physiotherapy intervention, in which the participants act as their own controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Individually tailored physiotherapy; cognitive behavioral intervention (Experimental): The intervention is offered in accordance with the Neck Pain Guidelines, with a focus on influencing dysfunctional illness perceptions and dysfunctional movement/ pain behavior.
  Interventions: Behavioral: Cognitive behavioral intervention

INTERVENTIONS:
Behavioral: Cognitive behavioral intervention — Individually tailored physiotherapy that fits within the guideline non-specific neck pain (KNGF, 2016) with a focus on influencing dysfunctional illness perceptions and dysfunctional movement/ pain behavior, by means of communication, body awareness exercises, functional movements and exposure techniques. Tools are supplied to create an appropriate explanatory model for the pain, for functional movement behavior and active coping in a patient's daily lives.

SUMMARY:
The aim of this study is to explore and evaluate the effects of an individually tailored intervention focusing on influencing dysfunctional illness perceptions and dysfunctional movement/pain behavior in patients with non-specific neck pain.

DETAILED DESCRIPTION:
Introduction:

Worldwide, neck pain is the 3th most common disorder that interferes with people's daily functioning. Many people with neck pain consult a physical therapist because of their pain, however treatment effects are small. Recent studies in a broader group of people with musculoskeletal pain show that physical therapy interventions tailored to individual risk profiles for chronicity are more effective. Considering the importance of psychological prognostic factors in neck pain it is hypothesized that influencing dysfunctional cognitions and negative emotions affects the way people cope with their pain and therefore can influence their self-perceived health condition in a positive way.

Research questions:

1. How does an individually tailored intervention that focuses on influencing dysfunctional illness perceptions and dysfunctional movement/ pain behavior change people's illness perceptions, the way they cope with their pain, their self-perceived health condition and to what do these people attribute this change?
2. Do changes in specific illness perceptions (i.e. cognitions and emotions measured by the IPQ-k and FABQ-pa) mediate the effect of an individually tailored physiotherapy cognitive behavioral intervention measured by the Global Perceived Effect, Self-efficacy (PSEQ), Functioning (PSFS) and Pain (NPRS).

Design:

In this study a Single Subject Experimental Design (SSED) is applied with a baseline phase (duration two weeks), an intervention phase with 5-7 treatment consultations (offered once a week) and a follow up (3 months after the last consultation).

During the baseline phase, a qualitative assessment of the illness perceptions, the way people cope with pain and their self-perceived health condition, is carried out through a semi-structured interview. A second interview is carried out after the treatment phase (in the week after the last treatment consultation) to explore changes in (1) the illness perceptions, (2) the way people cope with pain, (3) their self-perceived health condition and to explore to what these participants attribute a change in their perceived health condition.

The quantitative part of the study is used to investigate whether influencing illness perceptions (measured by the B-IPQ and the FABQ-pa) is a mediating factor for the treatment effect (i.e. self-perceived effect measured by the GPE scale, self-efficacy (PSEQ), functioning (PSFS) and pain (NPRS)). Outcome measurements in this quantitative part of the study will be performed two times a week during the baseline phase and the intervention phase. The last measurement in the intervention phase will be performed in the week after the treatment is completed (depending on the individual situation after 5-7 weeks of consultations). A follow-up measurement will be performed 3 months after the last treatment consultation.

Participants:

People with non-specific neck pain and a middle or high risk profile for chronicity (i.e. a score of ≥ 4 on the Start Neck Tool) are the target group for this study.

Procedure:

The study will be conducted in collaboration with 11 local physiotherapy clinics in primary health care. People with non-specific neck pain will be recruited via information on the website or social media channels of the physical therapy practices, via posters in the waiting room, via the secretary upon registration and via the physical therapist after the (regular) screening. After being screened by a physical therapist and when fulfilling the inclusion and exclusion criteria, information is given about the study. When willing to participate and after reading the information letter and signing the informed consent, patients will be included in the study. Their decision on participating in the study will not have consequences for their treatment. From enrollment, the participants will fill in the baseline measurements on the outcome variables twice a week and contact the researcher for making an appointment for an interview. The interview, performed by the leading researcher, will take place half way the baseline period of two weeks. In this interview the participant's illness perceptions, how they cope with their neck pain and their self-perceived health condition will be explored. Two weeks after enrollment in the study the intervention will start. The intervention, with a total of 5 till 7 treatment consultations depending on the patient's needs, is offered once a week by a trained physical therapist. During this phase, the self-reported outcome measures will be collected twice a week using questionnaires. The data from these questionnaires will be used to tailor the intervention. Within a week of completing the intervention, the researcher will be contacted and a second interview will take place. In addition to a further exploration of the participant's illness perceptions, how they cope with their pain and their self-perceived health condition at the end of the intervention, it is also evaluated to what the participant attributes a possible change in the perceived health condition and what the role of the intervention has been. Three months after the last treatment consultation, a follow up measurement will be conducted by completing a questionnaire on the aforementioned outcome variables.

Intervention:

The intervention consists of individually tailored physiotherapy that fits within the guideline non-specific neck pain (KNGF, 2016), with a focus on influencing dysfunctional illness perceptions and movement/pain behavior by means of communication, body awareness exercises, functional movements and exposure techniques. Depending on the patient's needs, 5-7 treatment consultations will be offered with a frequency of once a week. The intervention will be delivered by a trained physical therapist with specific interests in a cognitive-behavioral approach within a biopsychosocial model. The aim of the intervention is to influence dysfunctional beliefs and negative emotions to increase their self-perceived health condition and confidence in carrying out specific activities despite their pain and fulfill the patient's individually formulated goals.

Analyses:

This mixed method multiple case design implies the study of the clinical progress in an experimental set up by both a qualitative evaluation and frequent measurements of several quantitative outcome variables in a small sample of participants during a pre-intervention phase (A), an intervention phase (B) and an intervention withdrawal phase (A').

Qualitative analyses: Within the qualitative part of the study a content analysis will be conducted using the inductive analytical approach. The following steps will be taken: 1. Open coding (identifying domains and topics guided by the research questions) 2. Development of categories into a framework 3. Interpretation of the raw data 4. Discussion about the interpretations.

Quantitative analyses: Within the quantitative part of the study the participants are seen as single systems in the analyses and they act as their own controls. Repeated measures will be used to verify whether changes in specific illness perceptions (i.e. cognitions and emotions measured by the IPQ-k and FABQ-pa) mediates the effect of an individually tailored physiotherapy cognitive behavioral intervention on Global Perceived Effect, Self-efficacy, Functioning and Pain. Furthermore this quantitative research will be used to validate the data and interpretations from the interviews (i.e. to check whether 'the story people tell' corresponds to more objective markers (triangulation)).

Complementary Data:

Complementary data that will be collected within the project are the characteristics of the participating physical therapists (i.e. gender, age, work experience and specializations) and treatment related data (i.e. the number of physiotherapy sessions, the focus area within a session and the use of specific tools).

ELIGIBILITY:
Inclusion Criteria:

* Neck pain with no signs of major pathology, but with interference on daily activities (i.e., neck pain Grade II
* Aged 18-65
* The neck pain is present for a minimum of 2 weeks and pain and/or disability continues or increases
* A minimum score of 4 on the Start Neck Tool
* Good command of the Dutch language

Exclusion Criteria:

* Neck pain with neurological signs (i.e., neck pain Grade III) or neck pain with signs of serious pathology (i.e., neck pain Grade IV)
* Psychiatric disorders
* Surgery in the neck-arm area (< 3 months) and/or an acute mechanical trauma (< 3 weeks) in history

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-04-03 (Actual)

PRIMARY OUTCOMES:
Change in qualitative outcomes on illness perceptions, coping, self-perceived health condition and evaluating treatment: two semi-structured interviews will be conducted | Change in illness perceptions, coping and health condition from week 1 (i.e. mid-baseline, one week before the start of the intervention phase) till a week after the end of the intervention (i.e. week 9 or 10)
  An exploration of changes in (1) illness perceptions, (2) how people cope with their neck pain, (3) their perceived health condition and (4) to what they attribute a change in their perceived health condition during individually tailored physiotherapy treatment
Change in Global Perceived Effect Scale (GPES) (7-points Likert scale) (Quantitative outcome measurement) | Immediately after the first treatment consultation (week 3) and the second (week 4), third (week 5), fourth (week 6) and the fifth (+sixth/seventh) consultation (week 7 (+8/9) and at 3 months after the last consultation (i.e. follow up week 19/21)
  The GPES is a self-administered measure used to investigate the participant's perception of effect from the intervention they received. The GPES is scored on a seven-level Likert scale (1=Very much improved, 2=Much improved, 3=A little improved, 4=No change, 5=A little deterioration, 6=Much deterioration, 7=Very much deterioration)

SECONDARY OUTCOMES:
Pain Self-Efficacy (assessed by the Pain Self-Efficacy Questionnaire (PSEQ-2 / PSEQ-4)) | Scored twice a week from enrollment to the last (i.e. fifth, sixth or seventh) treatment consultation and three months after de last consultation (regardless of whether this was the 5th, 6th or 7th consultation)
  The Pain Self-Efficacy Questionnaire (PSEQ-2 / PSEQ-4) is used to assess participants' level of confidence in performing activities despite their pain. 5 Items scored on a 0 - 6 Scale (0=not at all confident, 6 = completely confident).
Functional Disability (assessed by the Patient Specific Functional Scale (PSFS)) | Scored twice a week from enrollment to the last (i.e. fifth, sixth or seventh) treatment consultation and three months after de last consultation
  The Patient Specific Functional Scale (PSFS) is used to identify and measure changes in the participant's ability to perform up to two self-selected activities regarded as important by them. Ability levels scored 0 - 10 (0= able to perform activity at the same level as before injury or problem, 10 = unable to perform activity)
Average Pain Intensity (assessed by the Numeric Pain Rating Scale (NPRS)) | Scored twice a week from enrollment to the last (i.e. fifth, sixth or seventh) treatment consultation and three months after de last consultation
  The average pain intensity within the last week (7 days) is measured by a 11-point numeric pain rating scale (NPRS) ranging from 0='no pain' to 10='worst pain imaginable'.

OTHER OUTCOMES:
Illness Perceptions (assessed by the Brief Illness Perception Questionnaire (B-IPQ)) | Scored twice a week from enrollment to the last (i.e. fifth, sixth or seventh) treatment consultation and three months after de last consultation
  The Brief Illness Perception Questionnaire (B-IPQ) is used to evaluate participants' illness perceptions. 8 Items scored on a 0-10 scale. After reversing items 3, 4 and 7 a higher score represents more dysfunctional beliefs. No sum-score can be measured, so each item will be evaluated separately.
Fear avoidance Beliefs (assessed by the Fear Avoidance Belief Questionnaire- physical activity subscale) | Scored twice a week from enrollment to the last (i.e. fifth, sixth or seventh) treatment consultation and three months after de last consultation
  The Fear Avoidance Belief Questionnaire (FABQ)-physical activity subscale is used to measure participant's beliefs about how physical activity affect their neck pain. 4 items scored on a 0 - 6 scale (0=completely disagree, 6=completely agree). A higher score represents more dysfunctional beliefs.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Coppieters, Prof., Study Chair — VU Amsterdam, The Netherlands; Griffith University, Australia
Locations (1):
- Rotterdam University of Applied Sciences, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Data available to share include the quantitative data collected during the trial, after deidentification.
Supporting Information: ICF
Time Frame: Informed Consent Form (ICF) - English language version will be available from the start of the study [1-11-2021] till the end of the study [expected date:1-11-2022]
Access Criteria: Investigators whose proposed use of the data has been approved by the national ethics committee. Proposals should be directed to the principal investigator. To gain access, data requestors will need to sign a data access agreement.

DOCUMENTS (1):
  • Informed Consent Form (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT05127603/ICF_000.pdf